CLINICAL TRIAL: NCT01033357
Title: A Long Term Safety Study of the Vascular Wrap(TM) Paclitaxel-Eluting Mesh After Surgical Implantation With the Lifespan® Graft in the Upper Extremity for Hemodialysis Vascular Access
Brief Title: Safety Study of the Vascular Wrap Paclitaxel-Eluting Mesh for Hemodialysis Vascular Access
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Imbalance in the # graft infections between the tx's (graft vs. graft + wrap)
Sponsor: Angiotech Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 014-VWAV07
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: End Stage Renal Failure on Dialysis; Hyperplasia
Keywords: dialysis; hemodialysis; neointimal hyperplasia
MeSH Terms: conditions — Hyperplasia | interventions — Transplantation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Graft, Vascular Wrap (Active Comparator): Lifespan® ePTFE Vascular Graft and Vascular Wrap Paclitaxel-Eluting Mesh (0.9 µg/mm2 paclitaxel)
  Interventions: Device: Graft, Vascular Wrap
- Graft (Placebo Comparator): Lifespan® ePTFE Vascular Graft Only
  Interventions: Device: Lifespan® ePTFE Vascular Graft Only

INTERVENTIONS:
Device: Graft, Vascular Wrap — Lifespan® ePTFE Vascular Graft and Vascular Wrap Paclitaxel-Eluting Mesh (0.9 µg/mm2 paclitaxel)
  Other Names: Vascular Wrap
  Arms: Graft, Vascular Wrap
Device: Lifespan® ePTFE Vascular Graft Only — Vascular Graft only
  Arms: Graft

SUMMARY:
The purpose of this study is to determine whether the long term use of the experimental Vascular Wrap(TM) Paclitaxel-Eluting Mesh is safe in the treatment of subjects needing hemodialysis access (via an expanded polytetrafluoroethylene (ePTFE) graft).

DETAILED DESCRIPTION:
The primary objective of this study is to determine long term safety of the Lifespan® ePTFE Vascular Graft and Vascular Wrap(TM) Paclitaxel-Eluting Mesh in comparison to the Lifespan® graft alone.

ELIGIBILITY:
Inclusion Criteria: To be considered for enrollment, subjects must:

* have been randomized in protocol 012-VWAV06;
* have signed and dated an IRB-approved written informed consent to participate in 012-VWAV06 as well as this study;
* be willing to comply with all aspects of the evaluation schedule over a period of 60 months post device insertion;
* allow representatives of the sponsor, designated Clinical Research Organization (CRO), Institutional Review Board (IRB), the Ethics Committee, and U.S. Food and Drug Administration (FDA) to review his/her relevant medical records.

Exclusion Criteria:

* Subjects who withdrew or were withdrawn from study 012-VWAV06.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2008-03; Primary Completion 2010-03 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Nature and incidence of Adverse Events between treatment groups clinical difference in product-related adverse events | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Rui Avelar, M.D., Study Chair — Angiotech Pharmaceuticals
Locations (30):
- United States (30):
  - Ladenheim, Inc., Fresno, California
  - Centinela Hospital, Inglewood, California
  - National Institute of Clinical Research, Los Angeles, California
  - USC CVTI - Healthcare Consultation II, Los Angeles, California
  - UCSD Medical Center, San Diego, California
  - Southern California Permanente Medical Group, San Diego, California
  - San Francisco VA Medical Center, San Francisco, California
  - Florida Research Network, LLC, Gainsville, Florida
  - Jacksonville Center for Clincal Research, Jacksonville, Florida
  - Discovery Medical Research Group, Ocala, Florida
  - Baptist Hospital, Pensacola, Florida
  - University of South Florida- Research Foundation, Tampa, Florida
  - Cardiothoracic and Vascular Surgery Associates, Macon, Georgia
  - Renal Care Associates, Peoria, Illinois
  - Southern Illinois University, Springfield, Illinois
  - Indiana University, Indianapolis, Indiana
  - Washington County Hospital Association, Hagerstown, Maryland
  - Michigan Vascular Research Center, Flint, Michigan
  - Thoracic and Cardiovascular Healthcare Foundation, Lansing, Michigan
  - Nephrology Associates P. C., Flushing, New York
  - St. Luke's Roosevelt Hospital Center, New York, New York
  - BRANY - Montefiore Medical Center, The Bronx, New York
  - Rex Healthcare, Raleigh, North Carolina
  - Clinical Research of Winston-Salem, Inc., Winston-Salem, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University of Toledo, Toledo, Ohio
  - Health First Medical Group, Fort Worth, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - Peripheral Vascular Associates, San Antonio, Texas
  - The Wisconsin Heart Hospital, Wauwatosa, Wisconsin